CLINICAL TRIAL: NCT02144402
Title: Growth of Healthy Term Infants Fed Formula Containing DHA-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Accelovance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-1069
Record Dates: First submitted 2014-05-16; First posted 2014-05-22 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Growth; Tolerance; Infant Development
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- infant formula with DHASCO (Active Comparator): standard infant formula with docosahexaenoic acid (DHA)
  Interventions: Other: infant formula with DHASCO
- infant formula with DHASCO-B (Experimental): standard infant formula with DHA-B
  Interventions: Other: infant formula with DHASCO-B

INTERVENTIONS:
Other: infant formula with DHASCO
  Arms: infant formula with DHASCO
Other: infant formula with DHASCO-B
  Arms: infant formula with DHASCO-B

SUMMARY:
The primary objective is to determine if the weight gain of healthy term infants fed a commercially available term infant formula supplemented with DHASCO® is similar to that of infants fed the same formula supplemented with a new product, DHASCO®-B.

ELIGIBILITY:
Inclusion Criteria:

* full term infant (gestational age 37-42 weeks)
* birth weight > or equal to 2500 g
* singleton infant < or equal to 14 days of age in good health
* parent must be >21 years of age
* parental consent

Exclusion Criteria:

* congenital malformation or genetic disorder
* metabolic anomalies
* maternal infectious diseases, alcoholism, substance abuse
* mothers with gestational diabetes
* participation in another clinical study

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
weight gain (gm/day) | through day of life 120
  gm/day -calculated from the weight measured at enrollment subtracted from the weight measured at DOL 120 visit, divided by the number of days between the actual visits.

SECONDARY OUTCOMES:
length (cm) | through day of life 120
  Length in cm
head circumference (cm) | through day of life 120
  head circumference (cm)
fatty acid levels (wgt %) | at day of life 120
  red blood cell (RBC) levels of omega-3 and omega-6 fatty acids (wgt %) in a sample subset
Formula intake and tolerance | Day of life 30 and 120
  assessed by analyzing three-day dietary intake and tolerance forms

OTHER OUTCOMES:
adverse events | through day of life 120
  AEs collected throughout the study

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Claude Ashley, MD, Dothan, Alabama
  - JBRKIDS, Jonesboro, Arkansas
  - Norwich Pediatric, Norwich, Connecticut
  - Score Physician Alliance, St. Petersburg, Florida
  - Atlantic Clinical Research, Wellington, Florida
  - Pedia Research, Newburgh, Indiana
  - Heartland Research, Wichita, Kansas
  - Stephen Kasparian, Fall River, Massachusetts
  - MCHRI, Lincoln, Nebraska
  - Ohio Pediatric Research, Dayton, Ohio